CLINICAL TRIAL: NCT02023749
Title: Effects of Nut Consumption on Metabolic Syndrome in Korean Adults - A Randomized Controlled Dietary Intervention Trial
Brief Title: Effects of Nut Consumption on Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Food and Drug Safety, Korea (Other Government)
Responsible Party: Principal Investigator, Nan Hee Kim, Prof, Korea University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12161MFDS118; 12161MFDS118 (Other Grant/Funding Number: Ministry of Food and Drug Safety)
Record Dates: First submitted 2013-12-17; First posted 2013-12-30 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Metabolic Syndrome
Keywords: nuts; metabolic syndrome; lipid profile; inflammation; oxidative stress; endothelial function
MeSH Terms: conditions — Metabolic Syndrome; Inflammation

ARMS (2):
- Nut group (Active Comparator): Subjects were supplemented with 30 g of mixed nuts including walnuts, peanuts, and pine nuts for 6 weeks
  Interventions: Dietary Supplement: Nut group
- Control group (No Intervention): Control group maintained their usual diet without nut supplement

INTERVENTIONS:
Dietary Supplement: Nut group
  Arms: Nut group

SUMMARY:
This study aimed to investigate the effects of nut consumption on metabolic parameters and biomarkers related to inflammation, oxidative stress, and endothelial function in Korean adults with metabolic syndrome.

DETAILED DESCRIPTION:
A randomized, controlled, parallel, dietary intervention study was designed. Subjects with metabolic syndrome and body mass index ≥23 kg/m2 were randomized to the Nut group, which were supplemented with 30 g of mixed nuts including walnuts, peanuts, and pine nuts for 6 weeks; or allocated to the Control group. Metabolic markers were evaluated at baseline and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were enrolled if their body mass index (BMI) was ≥23 kg/m2 and they met the criteria for metabolic syndrome.

Exclusion Criteria:

* Subjects were excluded if they had a nut allergy, peptic disorder, a history of cancer or cardiovascular disease including coronary artery disease, heart valve disease, or stroke, or established chronic diseases such as chronic renal insufficiency or cirrhosis. Subjects were also excluded if they:1) were receiving treatment with hypoglycemic agents for diabetes or had HbA1c >7%; 2) were receiving corticosteroid treatment; 3) had started antihypertensive or lipid-lowering agents, or changed their doses within the previous month; 4) had a weight change ≥5 % of body weight during the three months prior to the study; 5) were pregnant; or 6) were regular nut consumers (>15g/day of nuts at least three times a week).

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
metabolic parameters | 6 weeks
  lipid profiles, body mass index, waist circumference, blood pressure, fasting glucose, insulin, hemoglobin A1c and homeostasis model assessment of insulin resistance
inflammation markers | 6 weeks
  white blood cell count, high-sensitive C-reactive protein, Interleukin-6, adiponectin, serum and urine malondialdehyde, oxidized low-density lipoprotein, vascular cell adhesion molecule (VCAM) and intercellular adhesion molecule (ICAM)
Endo-peripheral artery tonometry (EndoPAT) index | 6 weeks
  EndoPAT index was assessed to evaluate endothelial function by using a finger plethysmograph based on non-invasive peripheral artery tonometry.

CONTACTS AND LOCATIONS:
Overall Officials: Nan Hee Kim, Prof, Principal Investigator — Department of Endocrinology and Metabolism, Korea University Ansan Hospital
Locations (1):
- Department of Endocrinology and Metabolism, Korea University Ansan Hospital, Ansan-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Lee YJ, Nam GE, Seo JA, Yoon T, Seo I, Lee JH, Im D, Bahn KN, Jeong SA, Kang TS, Ahn JH, Kim DH, Kim NH. Nut consumption has favorable effects on lipid profiles of Korean women with metabolic syndrome. Nutr Res. 2014 Sep;34(9):814-20. doi: 10.1016/j.nutres.2014.08.011. Epub 2014 Aug 30. PMID 25238912